CLINICAL TRIAL: NCT04838041
Title: Protocol Number: HJKC3-0003. Treatment Free Remission After Asciminib Based Therapy in Chronic Phase Chronic Myeloid Leukemia (CP-CML) Patients Who Relapsed After a Prior Attempt at TKI Discontinuation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: H. Jean Khoury Cure CML Consortium (Other)
Responsible Party: Principal Investigator, Ehab L Atallah, Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00040685
Record Dates: First submitted 2021-03-26; First posted 2021-04-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Phase Chronic Myelogenous Leukemia
Keywords: chronic myelogenous leukemia; treatment-free remission; tyrosine kinase inhibitors; H. Jean Khoury Cure CML Consortium; Asciminib
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib; Imatinib Mesylate; nilotinib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Asciminib 40 mg PO daily plus imatinib (maximum dose of 400 mg PO once daily) (Experimental): All eligible patients will begin asciminib plus/minus TKI on cycle 1 day 1 of the consolidation phase. They will continue therapy for a total of 12 cycles (minimum of 12 months). Each cycle will be ~28 days. At the end of 12 cycles, asciminib plus/minus TKI will be discontinued in patients who continue to satisfy the requirements for TFR attempt.
  Interventions: Drug: Asciminib 40 MG; Drug: Imatinib
- Asciminib 40 mg twice daily plus nilotinib (maximum dose of 300 mg twice daily) (Experimental): All eligible patients will begin asciminib plus/minus TKI on cycle 1 day 1 of the consolidation phase. They will continue therapy for a total of 12 cycles (minimum of 12 months). Each cycle will be ~28 days. At the end of 12 cycles, asciminib plus/minus TKI will be discontinued in patients who continue to satisfy the requirements for TFR attempt.
  Interventions: Drug: Asciminib 40 MG Twice Daily; Drug: Nilotinib
- Asciminib 80 mg daily plus dasatinib (maximum dose of 100 mg PO once daily) (Experimental): All eligible patients will begin asciminib plus/minus TKI on cycle 1 day 1 of the consolidation phase. They will continue therapy for a total of 12 cycles (minimum of 12 months). Each cycle will be ~28 days. At the end of 12 cycles, asciminib plus/minus TKI will be discontinued in patients who continue to satisfy the requirements for TFR attempt.
  Interventions: Drug: Asciminib 80 MG daily; Drug: Dasatinib
- Asciminib 80 mg PO daily taken alone (Experimental): All eligible patients will begin asciminib plus/minus TKI on cycle 1 day 1 of the consolidation phase. They will continue therapy for a total of 12 cycles (minimum of 12 months). Each cycle will be ~28 days. At the end of 12 cycles, asciminib plus/minus TKI will be discontinued in patients who continue to satisfy the requirements for TFR attempt.
  Interventions: Drug: Asciminib 80 MG daily

INTERVENTIONS:
Drug: Asciminib 40 MG — 40 mg by mouth (PO) when used with imatinib.
  Other Names: ABL001
  Arms: Asciminib 40 mg PO daily plus imatinib (maximum dose of 400 mg PO once daily)
Drug: Asciminib 40 MG Twice Daily — 40 mg twice daily when used with nilotinib.
  Other Names: ABL001
  Arms: Asciminib 40 mg twice daily plus nilotinib (maximum dose of 300 mg twice daily)
Drug: Asciminib 80 MG daily — 80 mg daily when used with dasatinib or taken alone.
  Other Names: ABL001
  Arms: Asciminib 80 mg PO daily taken alone; Asciminib 80 mg daily plus dasatinib (maximum dose of 100 mg PO once daily)
Drug: Imatinib — Maximum dose of 400 mg PO once daily.
  Other Names: Gleevec
  Arms: Asciminib 40 mg PO daily plus imatinib (maximum dose of 400 mg PO once daily)
Drug: Nilotinib — Maximum dose of 300 mg twice daily.
  Other Names: TASIGNA
  Arms: Asciminib 40 mg twice daily plus nilotinib (maximum dose of 300 mg twice daily)
Drug: Dasatinib — Maximum dose of 100 mg PO once daily.
  Other Names: Sprycel
  Arms: Asciminib 80 mg daily plus dasatinib (maximum dose of 100 mg PO once daily)

SUMMARY:
This is a single arm phase II study that will enroll a minimum of 47 subjects with a maximum of 51. All patients will have a confirmed diagnosis of chronic phase chronic myeloid Leukemia and must have previously attempted to discontinue Tyrosine Kinase inhibitors (TKI). All patients must have restarted the same TKI they were on prior to discontinuation at the time of relapse in order to be eligible for this trial.

DETAILED DESCRIPTION:
All eligible patients will begin asciminib plus/minus TKI on cycle 1 day 1 of the consolidation phase. They will continue therapy for a total of 12 cycles (minimum of 12 months). Each cycle will be ~28 days. At the end of 12 cycles, asciminib plus/minus TKI will be discontinued in patients who continue to satisfy the requirements for TFR attempt. The primary endpoint of this study is the 12-month 'second' TFR rate after completion of 12 cycles of asciminib based therapy. Patients will remain in the TFR phase of the study for up to three years and will have central PCR testing during the first two years. PCR testing will continue locally thereafter. Therefore, the total duration of the subject participation trial will be approximately five years (one year on consolidation phase + three years in the TFR phase + one year of long-term follow-up post TFR or early discontinuation.

ELIGIBILITY:
Eligibility for Consolidation Treatment Phase

Inclusion Criteria:

1. Age ≥18 years old.
2. Willing and able to give informed consent.
3. Diagnosed with chronic myelogenous leukemia (CML) in chronic phase without BCR::ABL1 ^T315I and have either the b3a2 (e14a2) or b2a2 (e13a2) variants that give rise to the p210 BCR::ABL1 protein. Subtype classification whether b3a2 (e14a2) or b2a2 (e13a2) is not required for study eligibility.
4. Must have a documented history of attempting only one prior TKI discontinuation under the guidance of a treating physician. TKI includes dasatinib, imatinib or nilotinib.
5. Must have met all the following criteria prior to first attempt to discontinue their TKI:

   * Stable molecular response (MR4; < 0.01% IS) for > 2 years (with allowance for a two-week variance), as documented on at least four tests, performed at least three months apart (e.g., If a patient has had >4 PCR tests performed during the two years leading up to their initial TKI discontinuation, any value between 0.01 and 0.05% IS is considered a stable result, however, at least four tests must be < 0.01% IS. If any results are >0.05% IS, tests must have been repeated within one month and be less than 0.01% IS and stable.
   * Treatment with one of the following FDA approved TKIs; imatinib, dasatinib, nilotinib at any dose for a minimum of approximately three years (allowance of a four-week variance) prior to discontinuing TKIs.
   * Has been on any number of TKIs, but has not been resistant to any TKI (changes made for intolerance are allowed).
6. Must have relapsed (defined as loss of major molecular response (MMR), RQ-PCR for BCR::ABL1 >0.1% IS after first attempted TKI discontinuation.
7. After first failed TFR attempt, must have a minimum duration of one year of retreatment with TKI, and must plan to remain on that TKI or switch to asciminib for a minimum of 12 months during the consolidation treatment phase.
8. Current TKI must be the same as the TKI being taken prior to the initial TFR attempt (e.g., if patient is on imatinib prior to first TFR attempt, they should be on imatinib at time of enrollment on this study).
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-3.
10. Must have a RQ-PCR for BCR::ABL1 < 0.0032% IS (MR4.5) reported by the trial designated central lab at the time of study enrollment.
11. Lipase ≤ 1.5 x upper limit of normal (ULN). For lipase > ULN - ≤ 1.5 x ULN, value should be considered not clinically significant and not associated with risk factors for acute pancreatitis.
12. eGFR ≥ 30 mL/min as calculated using the 2021 chronic kidney disease epidemiology (CKD-EPI) creatinine equation (https://www.kidney.org/professionals/kdoqi/gfr_calculator)
13. Female patients must meet one of the following:

    * Postmenopausal for at least one year before the screening visit,
    * Surgically sterile
    * If they are of childbearing potential, agree to practice two effective methods of contraception from the time of signing of the informed consent form through 90 days after the last dose of study drug,
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
14. Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:

    * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose.
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable.
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

1. History of accelerated or blast phase CML.
2. A second malignancy requiring active treatment.
3. History of recent (within 12 months) acute pancreatitis or chronic pancreatitis.
4. Subjects who have previously received treatment with asciminib.
5. Subjects with platelet (PLT) count < 100 × 109/L or an absolute neutrophil count (ANC) of < 1 × 109/L or hemoglobin < 8 g/dL.
6. Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≥3 times the institutional upper limit of normal.
7. Total bilirubin ≥ 1.5 times the institutional upper limit of normal (unless direct bilirubin is within normal limits).
8. Pregnant or lactating.
9. Unable to comply with lab appointment schedule and patient-reported outcome (PRO) assessments.
10. Another investigational drug within four weeks of enrollment.
11. Any serious medical or psychiatric illness that could, in the investigator's opinion, interfere with the completion of treatment according to this protocol.
12. Patient has undergone a prior allogeneic stem cell transplant.
13. Screening 12-lead electrocardiogram (ECG) showing a baseline corrected QT interval >480msec (patients with a pacemaker will still be eligible with QTc>500msec).
14. Known active hepatitis B infection.

Eligibility for TFR Phase:

1. Stable molecular response (MR4.5; < 0.0032% IS) documented on at least three tests (may include TFR phase screening PCR) by the trial designated lab, performed approximately three months apart while on consolidation phase.
2. TFR phase screening PCR RQ-PCR for BCR::ABL1 < 0.0032% IS (MR4.5) by the trial designated lab.
3. ECOG 0-3.
4. Completion of 12 cycles on the consolidation therapy phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
One-year "second" treatment-free remission. | 1 year after stopping treatment
  This will be measured by the number of subjects who achieve one-year treatment-free remission after 12 months of asciminib based therapy. These subjects have previously failed a first treatment free remission attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Atallah, MD, Principal Investigator — Medical College of Wisconsin; Michael J. Mauro, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - The Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No